CLINICAL TRIAL: NCT05417100
Title: Modulation of Post-operative Opioid Consumption and Pain by Intraoperative Methadone for Cancer Related Spinal Surgery - An Investigator Initiated Trial (IIT), Cluster Randomization Trial
Brief Title: Understanding How Methadone Treatment During Surgery Affects Pain Levels and the Need for Pain Medications After Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-015
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Spinal Surgery
Keywords: Methadone; Pain Levels; Pain Medications; 22-015
MeSH Terms: interventions — Methadone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methadone bolus during surgery (Active Comparator): Patients will be administered methadone 0.2 mg/kg (max 20 mg).
  Interventions: Drug: Methadone
- No Methadone during surgery (No Intervention): No Methadone during surgery

INTERVENTIONS:
Drug: Methadone — methadone 0.2 mg/kg IV.
  Arms: Methadone bolus during surgery

SUMMARY:
The researchers are doing this study to find out whether giving methadone during spinal surgery helps manage pain in the first 72 hours after surgery better than other standard pain medications. Participants' pain will be measured by how much pain is reported after surgery, and how much additional pain medication is needed to lower pain levels. The researchers will look at whether giving methadone during surgery reduces the need for other pain medications after surgery. In addition, the team will compare the effects of the two standard treatments- one with methadone and one without methadone to to evaluate which one works best.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (between 18-75 years of age) scheduled for extradural spine surgery with instrumentation (greater than or equal to two levels and including minimally invasive) of expected duration ≥ 2 hours
* Postoperative hospital stay expected to be ≥ 2 nights at the time of consent

Exclusion Criteria:

* Use of methadone currently or within the previous 6 weeks
* Drug misuse history (e.g., ketamine, cocaine, heroin, amphetamine, methamphetamine, MDMA, phencyclidine, lysergic acid, mescaline, psilocybin).
* Current use of opioid antagonist/partial antagonist (i.e. buprenorphine).
* Current or past diagnosis of a Major Psychiatric disorder (such as Schizophrenia, dementia, delirium).
* Patients with a BMI ≥ 36 kg/m2
* 2nd or 3rd degree heart block as assessed by preoperative EKG.
* QTc > 450 msec on preoperative EKG.
* Documentation of congestive heart failure and/or ejection fraction < 30% if recorded in the Pre-Operative Record.
* Contraindication to use of any analgesic medications listed in the ERAS pathways (acetaminophen, gabapentin, celecoxib, IV opioids).
* Any known hypersensitivity to methadone.
* Pregnant or breastfeeding.
* Abnormal liver function tests as related to the MSK guidelines for use of IV acetaminophen: ALT greater than 2 x Upper Limit of Normal (> 75 U/L)
* Serum Creatinine > 1.5 mg/dl
* Instrumented spine cases of less than 2 levels
* All non-instrumented spine cases
* All intradural tumor resections
* All "take backs" that occur within 72 hours of surgery (wound revisions, hematomas, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
opioid requirement in morphine equivalent | within 72 hours post-surgery
  To see if giving methadone during surgery reduces the need for other pain medications after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jess Brallier, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm